CLINICAL TRIAL: NCT02307500
Title: An Open-label Phase II Study of Regorafenib in Patients With Metastatic Solid Tumors Who Have Progressed After Standard Therapy - RESOUND
Brief Title: Regorafenib in Patients With Metastatic Solid Tumors Who Have Progressed After Standard Therapy
Acronym: RESOUND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2014-001
Record Dates: First submitted 2014-11-25; First posted 2014-12-04 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Pancreas Cancer; Ovarian Cancer; Melanoma; Sarcoma; Thymoma Type B3; Thymoma Type B2; Thymic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Ovarian Neoplasms; Melanoma; Sarcoma; Thymoma | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regorafenib (Experimental): Regorafenib 160 mg (40 mg tablets), po, every day for 3 weeks of every 4 week cycle
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — oral therapy
  Other Names: Stivarga

SUMMARY:
This is a single arm, single-stage, phase II trial to evaluate the activity of Regorafenib in patients with metastatic solid tumors (pancreatic cancer, ovarian cancer, melanoma, sarcoma, thymoma (type B2 - B3) and thymic carcinoma, who have progressed after standard therapy.

DETAILED DESCRIPTION:
Each tumour will be assessed by itself. Regorafenib 40 mg tablets will be used in the study. Subjects will receive 160 mg regorafenib po every day (qd) for 3 weeks of every 4 week cycle (i.e., 3 weeks on, 1 week off).

Subjects will continue on treatment until at least one of the following occurs (main criteria):

* Progressive Disease (PD) by radiological assessments or clinical progression
* Death
* Unacceptable toxicity
* Subject withdraws consent
* Treating physician determines discontinuation of treatment is in the subject's best interest
* Substantial non-compliance with the protocol

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Patients older then 18 years.
3. Locally advanced, recurrent or metastatic histologically confirmed malignancy refractory to available standard treatment, included Pancreatic cancer, Ovarian cancer, Melanoma, Sarcoma
4. At least one measurable lesion according to Response Evaluation Criteria In solid tumor
5. Eastern Cooperative Oncology Group Performance Status: 0-1
6. Life expectancy of at least 12 weeks
7. Adequate bone marrow, liver and renal function as assessed by the following laboratory : Hemoglobin > 9.0 g/dl Absolute neutrophil count > 1,500/mm3 Platelet count > 100,000/μl White blood cells >3.0 x 109/L Total bilirubin <1.5 times the upper limit of normal Alanine amino transferase and aspartate amino transferase <2.5 x upper limit of normal (<5 x upper limit of normal for patients with liver involvement) Serum creatinine <1.5 x upper limit of normal Alkaline phosphatase <2.5 x Upper Limit of Normal Prothrombin time / Partial prothrombin time <1.5 x Upper Limit of Normal Lipase ≤ 1.5 x the Upper Limit of Normal
8. Able to swallow and retain oral medication.
9. Estimated creatinine clearance > 30ml/min as calculated using the Cockcroft-Gault equation
10. Resolution of any toxic effects of prior therapy to NCI Common Terminology Criteria for Adverse Event, Version 4.0, grade ≤ 1 .
11. Women of childbearing potential and men must agree to use adequate contraception

Exclusion Criteria:

1. Prior treatment with regorafenib.
2. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study drug
3. Congestive heart failure >New York Heart Association class 2
4. Unstable angina), new-onset angina.Myocardial infarction less than 6 months before start of study drug
5. Myocardial infarction less than 6 months before start of study drug.
6. Cardiac arrhythmias requiring anti-arrhythmic therapy
7. Uncontrolled hypertension.
8. Pleural effusion or ascites that causes respiratory compromise
9. Ongoing infection > Grade 2
10. Known history of human immunodeficiency virus infection.
11. Active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy.
12. Subjects with seizure disorder requiring medication.
13. History of organ allograft. Subjects with evidence or history of any bleeding diathesis, irrespective of severity.
14. Any hemorrhage or bleeding event > Common Toxicity Criteria for Adverse Effects Grade 3
15. Arterial or venous thrombotic or embolic events within the 6 months before start of study medication
16. Known history or symptomatic metastatic brain or meningeal tumors
17. Suggestive or consistent with central nervous system disease
18. Renal failure requiring hemo-or peritoneal dialysis.
19. Dehydration Common Toxicity Criteria for Adverse Effects v. 4.0 Grade >1.
20. Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
21. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation.
22. Any illness or medical conditions that are unstable or could jeopardize the safety of the subject and his/her compliance in the study.
23. Interstitial lung disease with ongoing signs and symptoms
24. Persistent proteinuria of CTCAE Grade 3
25. Any malabsorption condition.
26. Concomitant participation or participation within the last 30 days in another clinical trial
27. Systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and hormonal therapy during this trial or within 4 weeks before starting to receive study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-12; Primary Completion 2017-12 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
activity of regorafenib screening, in terms of 2-months progression free survival rate | 2 months
  to evaluate activity of regorafenib, in terms of 2-months progression free survival rate

SECONDARY OUTCOMES:
prognosis in terms of progression-free survival | 36 months
  to explore the prognosis in terms of progression-free survival calculated from the first day of regorafenib treatment to the date of tumor progression or death, whichever occurs first.
overall survival (OS) | 36 months
  to explore overall survival (OS) measured from the first day of regorafenib treatment until the date of death from any cause or the date of the last contact, at which the patients will be censored
safety profile of regorafenib according to NCI-CTC v.3 | 3 months
  to assess the safety profile of regorafenib according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 3

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy

REFERENCES:
- [Background] Wilhelm SM, Dumas J, Adnane L, Lynch M, Carter CA, Schutz G, Thierauch KH, Zopf D. Regorafenib (BAY 73-4506): a new oral multikinase inhibitor of angiogenic, stromal and oncogenic receptor tyrosine kinases with potent preclinical antitumor activity. Int J Cancer. 2011 Jul 1;129(1):245-55. doi: 10.1002/ijc.25864. Epub 2011 Apr 22. PMID 21170960
- [Background] Carmeliet P, Jain RK. Angiogenesis in cancer and other diseases. Nature. 2000 Sep 14;407(6801):249-57. doi: 10.1038/35025220. PMID 11001068
- [Background] Ferrara N. Vascular endothelial growth factor as a target for anticancer therapy. Oncologist. 2004;9 Suppl 1:2-10. doi: 10.1634/theoncologist.9-suppl_1-2. PMID 15178810
- [Background] Fong GH, Rossant J, Gertsenstein M, Breitman ML. Role of the Flt-1 receptor tyrosine kinase in regulating the assembly of vascular endothelium. Nature. 1995 Jul 6;376(6535):66-70. doi: 10.1038/376066a0. PMID 7596436
- [Background] Shalaby F, Rossant J, Yamaguchi TP, Gertsenstein M, Wu XF, Breitman ML, Schuh AC. Failure of blood-island formation and vasculogenesis in Flk-1-deficient mice. Nature. 1995 Jul 6;376(6535):62-6. doi: 10.1038/376062a0. PMID 7596435
- [Background] Goodman VL, Rock EP, Dagher R, Ramchandani RP, Abraham S, Gobburu JV, Booth BP, Verbois SL, Morse DE, Liang CY, Chidambaram N, Jiang JX, Tang S, Mahjoob K, Justice R, Pazdur R. Approval summary: sunitinib for the treatment of imatinib refractory or intolerant gastrointestinal stromal tumors and advanced renal cell carcinoma. Clin Cancer Res. 2007 Mar 1;13(5):1367-73. doi: 10.1158/1078-0432.CCR-06-2328. PMID 17332278
- [Background] Amit L, Ben-Aharon I, Vidal L, Leibovici L, Stemmer S. The impact of Bevacizumab (Avastin) on survival in metastatic solid tumors--a meta-analysis and systematic review. PLoS One. 2013;8(1):e51780. doi: 10.1371/journal.pone.0051780. Epub 2013 Jan 22. PMID 23349675
- [Background] Yancopoulos GD, Davis S, Gale NW, Rudge JS, Wiegand SJ, Holash J. Vascular-specific growth factors and blood vessel formation. Nature. 2000 Sep 14;407(6801):242-8. doi: 10.1038/35025215. PMID 11001067
- [Background] Acevedo VD, Ittmann M, Spencer DM. Paths of FGFR-driven tumorigenesis. Cell Cycle. 2009 Feb 15;8(4):580-8. doi: 10.4161/cc.8.4.7657. Epub 2009 Feb 18. PMID 19182515
- [Background] Bergers G, Song S, Meyer-Morse N, Bergsland E, Hanahan D. Benefits of targeting both pericytes and endothelial cells in the tumor vasculature with kinase inhibitors. J Clin Invest. 2003 May;111(9):1287-95. doi: 10.1172/JCI17929. PMID 12727920
- [Background] Augustin HG, Koh GY, Thurston G, Alitalo K. Control of vascular morphogenesis and homeostasis through the angiopoietin-Tie system. Nat Rev Mol Cell Biol. 2009 Mar;10(3):165-77. doi: 10.1038/nrm2639. PMID 19234476
- [Background] Huang J, Bae JO, Tsai JP, Kadenhe-Chiweshe A, Papa J, Lee A, Zeng S, Kornfeld ZN, Ullner P, Zaghloul N, Ioffe E, Nandor S, Burova E, Holash J, Thurston G, Rudge J, Yancopoulos GD, Yamashiro DJ, Kandel JJ. Angiopoietin-1/Tie-2 activation contributes to vascular survival and tumor growth during VEGF blockade. Int J Oncol. 2009 Jan;34(1):79-87. PMID 19082480
- [Background] Bach F, Uddin FJ, Burke D. Angiopoietins in malignancy. Eur J Surg Oncol. 2007 Feb;33(1):7-15. doi: 10.1016/j.ejso.2006.07.015. Epub 2006 Sep 7. PMID 16962282
- [Background] Saito M, Watanabe J, Fujisawa T, Kamata Y, Nishimura Y, Arai T, Miyamoto T, Obokata A, Kuramoto H. Angiopoietin-1, 2 and Tie2 expressions in endometrial adenocarcinoma--the Ang2 dominant balance up-regulates tumor angiogenesis in the presence of VEGF. Eur J Gynaecol Oncol. 2006;27(2):129-34. PMID 16620053
- [Background] Szarvas T, Jager T, Totsch M, vom Dorp F, Kempkensteffen C, Kovalszky I, Romics I, Ergun S, Rubben H. Angiogenic switch of angiopietins-Tie2 system and its prognostic value in bladder cancer. Clin Cancer Res. 2008 Dec 15;14(24):8253-62. doi: 10.1158/1078-0432.CCR-08-0677. PMID 19088043
- [Background] Turner N, Grose R. Fibroblast growth factor signalling: from development to cancer. Nat Rev Cancer. 2010 Feb;10(2):116-29. doi: 10.1038/nrc2780. PMID 20094046
- [Background] Fletcher JA, Rubin BP. KIT mutations in GIST. Curr Opin Genet Dev. 2007 Feb;17(1):3-7. doi: 10.1016/j.gde.2006.12.010. Epub 2007 Jan 8. PMID 17208434
- [Background] Lanzi C, Cassinelli G, Nicolini V, Zunino F. Targeting RET for thyroid cancer therapy. Biochem Pharmacol. 2009 Feb 1;77(3):297-309. doi: 10.1016/j.bcp.2008.10.033. Epub 2008 Nov 6. PMID 19028457
- [Background] Marshall CJ. MAP kinase kinase kinase, MAP kinase kinase and MAP kinase. Curr Opin Genet Dev. 1994 Feb;4(1):82-9. doi: 10.1016/0959-437x(94)90095-7. PMID 8193545
- [Background] Herrera R, Sebolt-Leopold JS. Unraveling the complexities of the Raf/MAP kinase pathway for pharmacological intervention. Trends Mol Med. 2002;8(4 Suppl):S27-31. doi: 10.1016/s1471-4914(02)02307-9. PMID 11927284
- [Background] Ferrara N. VEGF and the quest for tumour angiogenesis factors. Nat Rev Cancer. 2002 Oct;2(10):795-803. doi: 10.1038/nrc909. PMID 12360282
- [Background] Sawyers CL. Finding the next Gleevec: FLT3 targeted kinase inhibitor therapy for acute myeloid leukemia. Cancer Cell. 2002 Jun;1(5):413-5. doi: 10.1016/s1535-6108(02)00080-6. PMID 12124170
- [Background] Heinrich MC, Blanke CD, Druker BJ, Corless CL. Inhibition of KIT tyrosine kinase activity: a novel molecular approach to the treatment of KIT-positive malignancies. J Clin Oncol. 2002 Mar 15;20(6):1692-703. doi: 10.1200/JCO.2002.20.6.1692. PMID 11896121
- [Background] Nikiforov YE. Thyroid carcinoma: molecular pathways and therapeutic targets. Mod Pathol. 2008 May;21 Suppl 2(Suppl 2):S37-43. doi: 10.1038/modpathol.2008.10. PMID 18437172
- [Background] Apperley JF, Gardembas M, Melo JV, Russell-Jones R, Bain BJ, Baxter EJ, Chase A, Chessells JM, Colombat M, Dearden CE, Dimitrijevic S, Mahon FX, Marin D, Nikolova Z, Olavarria E, Silberman S, Schultheis B, Cross NC, Goldman JM. Response to imatinib mesylate in patients with chronic myeloproliferative diseases with rearrangements of the platelet-derived growth factor receptor beta. N Engl J Med. 2002 Aug 15;347(7):481-7. doi: 10.1056/NEJMoa020150. PMID 12181402
- [Background] Mross K, Frost A, Steinbild S, Hedbom S, Buchert M, Fasol U, Unger C, Kratzschmar J, Heinig R, Boix O, Christensen O. A phase I dose-escalation study of regorafenib (BAY 73-4506), an inhibitor of oncogenic, angiogenic, and stromal kinases, in patients with advanced solid tumors. Clin Cancer Res. 2012 May 1;18(9):2658-67. doi: 10.1158/1078-0432.CCR-11-1900. Epub 2012 Mar 15. PMID 22421192
- [Background] Grothey A, Van Cutsem E, Sobrero A, Siena S, Falcone A, Ychou M, Humblet Y, Bouche O, Mineur L, Barone C, Adenis A, Tabernero J, Yoshino T, Lenz HJ, Goldberg RM, Sargent DJ, Cihon F, Cupit L, Wagner A, Laurent D; CORRECT Study Group. Regorafenib monotherapy for previously treated metastatic colorectal cancer (CORRECT): an international, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2013 Jan 26;381(9863):303-12. doi: 10.1016/S0140-6736(12)61900-X. Epub 2012 Nov 22. PMID 23177514
- [Derived] Marrari A, Bertuzzi A, Bozzarelli S, Gennaro N, Giordano L, Quagliuolo V, De Sanctis R, Sala S, Balzarini L, Santoro A. Activity of regorafenib in advanced pretreated soft tissue sarcoma: Results of a single-center phase II study. Medicine (Baltimore). 2020 Jun 26;99(26):e20719. doi: 10.1097/MD.0000000000020719. PMID 32590747
- [Derived] Bozzarelli S, Rimassa L, Giordano L, Sala S, Tronconi MC, Pressiani T, Smiroldo V, Prete MG, Spaggiari P, Personeni N, Santoro A. Regorafenib in patients with refractory metastatic pancreatic cancer: a Phase II study (RESOUND). Future Oncol. 2019 Dec;15(35):4009-4017. doi: 10.2217/fon-2019-0480. Epub 2019 Nov 20. PMID 31746632